CLINICAL TRIAL: NCT06705517
Title: Mediterranean Diet Effects on Parkinson's Disease (MED-PARK): a Randomized Controlled Trial
Brief Title: Mediterranean Diet Effects on Parkinson's Disease
Acronym: MED-PARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Associazione Parkinson Insubria (AsPI), Section of Varese (Unknown); University of Piemonte Orientale (Unknown); Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Franca Marino, Professor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MED-PARK
Record Dates: First submitted 2024-11-14; First posted 2024-11-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-03

CONDITIONS: Parkinson; Parkinson Disease; Parkinson Disease, Idiopathic; PARKINSON DISEASE (Disorder)
Keywords: Diet; Mediterranean Diet; Parkinson; Parkinson disease; MIND diet; plant based diet; unprocessed diet
MeSH Terms: conditions — Parkinson Disease | interventions — Diet, Mediterranean; Diet Therapy

STUDY DESIGN:
Intervention Model Description: This is an interventional, non-pharmacological, superiority, randomized, controlled, single-center, masked study with two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors, including the study neurologist and researchers analyzing biological samples, will be blinded to the allocation of the patients. Patients will be instructed to keep this information confidential during their neurological evaluations. Before data analysis, the dataset will be anonymized a second time to perform a blind data analysis, so also investigators will be partially blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (standard of care + MD) (Experimental): The intervention group will participate in a six-month program aimed at promoting adherence to the MD. At the start, participants will be given a physical booklet outlining foods to prioritize and avoid. They will also receive monthly recipes featuring seasonal ingredients. In addition, cooking classes will be offered, with caregiver involvement encouraged.
  Interventions: Behavioral: Mediterranean Diet
- Control group (standard of care) (No Intervention): The control group will be asked to maintain their current dietary habits and usual standard care. They will undergo the same routine examinations and check-ups as the intervention group.

INTERVENTIONS:
Behavioral: Mediterranean Diet — The MD emphasizes a plant-based approach, with a high consumption of vegetables, fruits, whole grains, legumes, and nuts, alongside moderate amounts of fish, seafood, and dairy, while limiting meat, particularly red and processed varieties. Olive oil serves as the main fat source in the diet. In the case of this study participants will also be instructed to limit dairy intake, that although traditionally part of the MD, might exacerbate disease symptomatology in PD patients, likely due to the urate lowering effect of dairy.
  Other Names: Dietary intervention
  Arms: Intervention group (standard of care + MD)

SUMMARY:
Currently, there are no disease-modifying treatments for Parkinson's disease (PD), the second most common neurodegenerative disorder worldwide, making it crucial to find interventions that can change the disease's trajectory. Epidemiological studies suggest that the Mediterranean diet (MD) is linked to improved motor and non-motor symptoms, slower disease progression, and lower mortality in PD patients. However, few interventional studies have explored this connection. This study assesses whether an MD can improve motor and non-motor symptoms in PD patients. Additionally, the study will examine the effects of the diet on a patient's quality of life, gastrointestinal symptomatology, adaptive immune system, fecal and nasal microbiome, and fecal and urinary metabolomics.

This is a randomized, controlled, non-pharmacological, single-center, masked trial with two parallel groups. It will evaluate the safety and efficacy of the MD on motor and non-motor symptoms reported by PD patients. Forty-four participants, aged 40-85, meeting the inclusion criteria will be enrolled and block-randomized into two groups: one maintaining their usual diet (control) and the other following a MD for six months (intervention).

The primary outcome is patient-reported symptoms, measured using the MDS-UPDRS I+II score.

Secondary outcomes include the analysis of adaptive immune system cells, nasal and fecal microbiome composition, and inflammatory and metabolic markers. Additional assessments include disease severity (MDS-UPDRS), non-motor symptoms (Non-Motor Symptoms Scale), participant well-being (36-Item Short Form Health Survey), gastrointestinal symptoms (Gastrointestinal Symptom Rating Scale and Patient Assessment of Constipation Quality of Life), and the intensity of dopaminergic therapy (levodopa equivalents). Evaluations will be performed at baseline and after six months.

DETAILED DESCRIPTION:
PD is a progressive neurodegenerative disorder marked by both motor and non-motor symptoms, leading to reduced quality of life and increased economic burden for patients and caregivers. Prior to diagnosis, patients often experience a prodromal phase characterized by symptoms such as anosmia, constipation, and sleep disturbances. PD is the second most common neurodegenerative disease globally and the fastest-growing, with an increasing prevalence since 1990.

The disease is linked to the buildup of α-synuclein in Lewy bodies within the brain and neuroinflammation caused by microglial activation. This process results in the degeneration of dopaminergic neurons in the substantia nigra, which is central to PD pathology. Recent research has highlighted the role of immune dysfunction in PD, with alterations observed in adaptive and innate immune responses. A reduction in specific T cells (e.g., CD4+ T cells, Th2, Th17, and T regulatory cells) and a shift towards a pro-inflammatory Th1 response have been associated with neuronal damage in PD. Moreover, aberrant α-synuclein may trigger an adaptive immune response, highlighting the relevance of the immune system as a potential therapeutic target.

Gut and nasal microbiota also appear to play a role in PD. Alterations in the gut microbiome, including changes in short-chain fatty acid-producing bacteria, have been observed in PD patients. Notably, increases in Lactobacillus, Akkermansia, and Bifidobacterium have been reported in the gut, while the Lachnospiraceae family and Faecalibacterium genus are reduced.

Moreover, although still unconfirmed, nasal microbiota may contribute to neurodegeneration by traveling through the olfactory and trigeminal pathways, possibly initiating or exacerbating brain inflammation.

Evidence suggests that specific dietary patterns may influence PD risk and progression. Foods like dairy are associated with an increased risk of PD, while coffee, nicotine-containing vegetables (e.g., peppers and tomatoes), and high consumption of vegetables, nuts, and fish may reduce symptomatology.

The MD, a plant-based diet rich in vegetables, fruits, whole grains, and healthy fats like olive oil, has been linked to numerous health benefits, including improved cognitive function, cardiovascular health, and a reduced risk of developing PD.

Studies show that a high-fiber diet can positively impact α-synuclein aggregation and microglial activation. Adherence to the MD may lower PD risk by up to 26%, slow disease progression, and improve both motor and non-motor symptoms. In contrast to pharmacological treatments, the MD has minimal side effects and could address several unmet needs in PD management, particularly in slowing disease progression and reducing comorbidities such as dementia.

This six-month randomized controlled trial aims to explore whether strict adherence to the MD can stabilize or slow the progression of motor and non-motor symptoms in PD patients. It will also investigate the impact of the MD on the immune system, gut and nasal microbiota, and fecal metabolomics, making it the first trial to assess these factors together. The study's primary goal is to determine the benefits of MD adherence on symptom management while also exploring correlations between immune function, microbiota composition, fecal and urinary metabolomics, and diet adherence levels.

ELIGIBILITY:
Inclusion Criteria:

1. PD diagnosis according to international guidelines;
2. Age between 40 and 85 years;
3. Naive to medication or with a stable dosage of anti-Parkinson's therapy for at least two weeks;
4. Hoehn & Yahr stage ≤3;
5. Normal independent feeding;
6. Ability to complete informed consent;
7. Willingness to maintain the usual diet in the period between T0 and T1;
8. Willingness to maintain the usual diet if randomized to the control group in the T1-T2 period;
9. Willingness to make changes in their diet to follow a Mediterranean diet if randomized to the intervention group in the T1-T2 period;
10. Willingness to fill out questionnaires;
11. Willingness to provide blood samples during the study collection periods;
12. Willingness to provide stool samples during the study collection periods;
13. Willingness to fast (without food or drink except water, tea or coffee) at least 12 hours before each sample collection;
14. Willingness to discontinue taking supplements, probiotics, herbal or high- dose vitamins or minerals that could impact inflammation during the period between T0 and T1 and for the duration of the study protocol;
15. No medical and/or social conditions that could interfere with participation in a six-month interventional study.

Exclusion Criteria:

1. Atypical or secondary parkinsonism;
2. Underweight (<18.5);
3. Obesity (BMI>30);
4. Pregnancy or suspected pregnancy;
5. Normal assisted nutrition;
6. Enteral nutrition;
7. Chronic autoimmune diseases;
8. Chronic use of immunosuppressive drugs in the past year;
9. Chronic use of cytotoxic cancer drugs in the past year;
10. Major abdominal surgeries;
11. Concurrent participation in other interventional studies;
12. Intentional change in diet after PD diagnosis.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) I+II | Baseline - 6 months
  The primary outcome of this study is the mean (final - baseline) change in disease severity between the control and intervention groups at the end of the intervention, which will be assessed using the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) I+II score. Part I of the scale (13 items) investigates non-motor aspects of the disease, whilst part II (13 items) refers to motor aspects. The MDS-UPDRS will be performed at baseline and after 6 months. The scores in each item vary from 0 (normal) to 4(severe), Higher the score, the more severe the condition or symptom.

SECONDARY OUTCOMES:
Immunophenotype | Baseline - 6 months
  Flow cytofluorimetric assay of the immunophenotype of circulating cells of the adaptive immune system will be performed. The investigated subpopulations include naïve/memory CD4+ and CD8+ T cells, CD4+ helper T subsets (Th1, Th2, and Th17), CD4+ regulatory T cells (conventional, naïve, and activated Treg), monocytes (classical, nonclassical, and intermediate), and Natural Killer (NK CD56 dim CD56 bright) cells.
Intestinal and Nasal microbiota | Baseline - 6 months
  In this study, the effect of the MD on the composition (taxonomy) and quantity of the intestinal and nasal microbiota will be evaluated.
  Both nasal and intestinal microbiota will be analyzed by sequencing the bacterial 16S rRNA gene, which will be amplified using universal bacterial primers to assess the composition and quantity of the intestinal and nasal microbiota. We will examine operational taxonomic units (OTUs) as well as alpha and beta diversity.
Fecal metabolites | Baseline - 6 months
  Exposure to phenolic compounds will be assessed by analyzing metabolites and catabolites of (poly)phenols in the collected fecal samples.
Urinary metabolites | Baseline - 6 months
  Exposure to phenolic compounds will be assessed by analyzing metabolites and catabolites of (poly)phenols in the collected urinary samples.
Non-Motor Symptom Scale (NMSS) | Baseline - 6 months
  The NMSS is a 30-item rater-based scale that assesses the severity and frequency of non-motor symptoms across nine dimensions. Total scores range from 0 to 360, with higher scores indicating greater symptom burden.
Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline - 6 months
  The MDS-UPDRS is a partly rater-based and partly patient-based questionnaire that assesses disease severity through 65 items divided into four domains: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination), and Part IV (motor complications). The MDS-UPDRS is designed to assess the presence and severity of clinically relevant problems in various domains. Scores range from 0 to 272, with higher scores indicating greater severity.
  The full MDS-UPDRS will be assessed by the study neurologist during in-person visits. For each domain of the MDS-UPDRS and for the total scores of the MDS-UPDRS within each of the two study arms, baseline and final scores will be collected for each patient and each domain.
GSRS (Gastrointestinal Symptom Rating Scale) | Baseline - 6 months
  The GSRS is a self-reported 15-item questionnaire that assesses the severity of gastrointestinal symptoms over the course of one week. It evaluates the severity of gastrointestinal symptoms across five domains: reflux, abdominal pain, indigestion, diarrhea, and constipation. Scores range from 1 to 7, with higher scores indicating greater symptom severity.
The Pac-QoL (Patient Assessment of Constipation Quality of Life) | Baseline - 6 months
  The Pac-QoL is a self-reported 28-item questionnaire assessing the quality of life-related to constipation over the past two weeks. The PAC-QOL measures the impact of constipation on quality of life across four domains: physical discomfort, psychosocial discomfort, worries/concerns, and satisfaction. Scores range from 0 to 4, with higher scores indicating greater negative impact and lower scores reflecting better quality of life
Diet adherence - MEDAS (Mediterranean Diet Adherence Screener) | Baseline - 6 months
  The MEDAS questionnaire is a self-reported 14-item questionnaire that investigates eating habits and will allow the measurement of adherence to the MD, diet modification, and effectiveness of the lifestyle intervention.
  The MEDAS assesses adherence to the Mediterranean diet through 14 items, each scored as 1 (criterion met) or 0 (not met). Total scores range from 0 to 14, with ≥9 indicating good adherence and <9 reflecting moderate or low adherence. Higher scores suggest better alignment with Mediterranean dietary patterns, often linked to improved health outcomes.
Quality of life - SF-36 (36-Item Short Form Health Survey) | Baseline - 6 months
  The SF-36 is a standardized tool for assessing health-related quality of life across eight domains. Each domain is scored on a scale from 0 to 100, with 0 representing the poorest health and 100 representing the best possible health. These domains evaluate various aspects of physical and mental health, including physical functioning, bodily pain, vitality, and mental well-being.
Body Mass Index (BMI) | Baseline - 6 months
  Height will be measured while standing without shoes. Weight will be recorded without footwear and in light clothing using a digital scale with a precision of 100 grams. BMI will be determined by dividing weight by the square of height, expressed in kilograms per square meter (kg/m²).
Waist circumference | Baseline - 6 months
  Waist circumference will be measured according to the WC-mid protocol, following World Health Organization recommendations
Daily Levodopa Equivalent Dose | Baseline - 6 months
  Levodopa equivalents will be calculated using the free platform EQUIDopa to assess the intensity of dopaminergic replacement therapy and facilitate the confrontation of different therapy schedules. Physicians will collect data during inpatient visits at baseline and after 6 months.
Complete blood count with formula | Baseline - 6 months
  Collect the data of complete blood count with formula from blood test
Total Cholesterol | Baseline - 6 months
  Collect the data of serum concentration of Total Cholesterol from blood test
HDL Cholesterol | Baseline - 6 months
  Collect the data of serum concentration of HDL Cholesterol from blood test
LDL Cholesterol | Baseline - 6 months
  Collect the data of serum concentration of LDL Cholesterol from blood test
Triglycerides | Baseline - 6 months
  Collect the data of serum Triglycerides levels from blood test
Glycemia | Baseline - 6 months
  Collect the data of glucose levels from blood test
GOT (transaminase) | Baseline - 6 months
  Collect the data of GOT from blood test
GPT (transaminase) | Baseline - 6 months
  Collect the data of GOT from blood test
Gamma-glutamyl transferase | Baseline - 6 months
  Collect the data of Ggt from blood test
Erythrocyte Sedimentation Rate | Baseline - 6 months
  Collect the data of erythrocyte Sedimentation Rate from blood test
Creatinine | Baseline - 6 months
  Collect the data on creatinine levels from blood test
Azotemia | Baseline - 6 months
  Collect the data on nitrogen-containing compounds from blood test
Uricemia | Baseline - 6 months
  Collect the data on uric acid levels from blood test

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cosentino, MD, PhD, Principal Investigator — Università degli studi dell Insubria; Franca Marino, M.Sc., PhD, Principal Investigator — Università degli studi dell Insubria; Elenamaria Pirovano, MD, Principal Investigator — Università degli studi dell Insubria
Locations (1):
- Centre for Research in Medical Pharmacology, Varese, Varese, Italy

IPD SHARING:
Plan to Share IPD: Yes
After publication, upon reasonable request, the anonymized dataset will be provided.
Supporting Information: Study Protocol, ICF
Time Frame: After the study conclusion and publication of results

REFERENCES:
- [Background] Kustrimovic N, Rasini E, Legnaro M, Bombelli R, Aleksic I, Blandini F, Comi C, Mauri M, Minafra B, Riboldazzi G, Sanchez-Guajardo V, Marino F, Cosentino M. Dopaminergic Receptors on CD4+ T Naive and Memory Lymphocytes Correlate with Motor Impairment in Patients with Parkinson's Disease. Sci Rep. 2016 Sep 22;6:33738. doi: 10.1038/srep33738. PMID 27652978
- [Background] Kustrimovic N, Comi C, Magistrelli L, Rasini E, Legnaro M, Bombelli R, Aleksic I, Blandini F, Minafra B, Riboldazzi G, Sturchio A, Mauri M, Bono G, Marino F, Cosentino M. Parkinson's disease patients have a complex phenotypic and functional Th1 bias: cross-sectional studies of CD4+ Th1/Th2/T17 and Treg in drug-naive and drug-treated patients. J Neuroinflammation. 2018 Jul 12;15(1):205. doi: 10.1186/s12974-018-1248-8. PMID 30001736
- [Derived] Pirovano E, Marino F, Rossi E, Gennari A, Rasini E, Uslenghi M, Figueira I, Iacoviello L, Ferrari M, Cosentino M. Modified Mediterranean diet effects on Parkinson's disease (MED-PARK): a single-centre randomised controlled trial protocol. BMJ Open. 2025 Oct 5;15(10):e101946. doi: 10.1136/bmjopen-2025-101946. PMID 41047258